CLINICAL TRIAL: NCT04790071
Title: Does Dry Needling Treatment Make an Extra Contribution to Conventional Treatment in Hemiplegic Shoulder Pain?
Brief Title: Dry Needling Treatment in Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kars State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Bagcier, Study Principal Investigator, Kars State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-KAEK-43-20-12
Record Dates: First submitted 2021-02-27; First posted 2021-03-10 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Hemiplegia; Shoulder Pain; Myofascial Pain
Keywords: Hemiplegic shoulder pain; Conventional treatment; Dry needling
MeSH Terms: conditions — Hemiplegia; Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Prospective randomised controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): It covers the classical physical therapy modalities that patients will take for shoulder pain.
  Interventions: Other: Conventional physical therapy
- Conventional therapy plus dry needling (Active Comparator): It covers the classical physical therapy modalities that patients will take for shoulder pain. It also refers to the dry needling treatment to be applied.
  Interventions: Other: Conventional physical therapy plus dry needling

INTERVENTIONS:
Other: Conventional physical therapy — Conventional physical therapy: The patients received physical therapy to the shoulder, transcutaneous electrical nerve stimulation, and stretching and strengthening exercises (5 days per week for three weeks in a total of 15 sessions).
  Arms: Conventional therapy
Other: Conventional physical therapy plus dry needling — Conventional physical therapy plus dry needling: The patients received physical therapy to the shoulder, including transcutaneous electrical nerve stimulation, stretching, and strengthening exercise (5 days per week for three weeks in a total of 15 sessions). And also, a total of 3 dry needling sessions were applied at 7-day intervals.
  Arms: Conventional therapy plus dry needling

SUMMARY:
To evaluate the efficacy of dry needling therapy on shoulder pain and upper extremity functions in hemiplegic patients.

DETAILED DESCRIPTION:
The myofascial trigger point is an overlooked issue in hemiplegic shoulder pain. Our aim in this study is to evaluate whether dry needling treatment contributes to the conventional treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in the study were aged between 30-60 years, with at least a 3-month history of hemorrhagic or ischemic stroke.

Exclusion Criteria:

* if they had severe difficulty in communication
* had received a corticosteroid injection within 3 months prior to enrollment
* had bleeding diathesis, a history of shoulder surgery
* a preexisting painful shoulder disorder, or had a cardiac pacemaker.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
Change in visual analog scale score | 3 months
  It grades pain of the patients between 0 and 10 points. Higher scores represent a worse outcome
Change in range of motion | 3 months
  Shoulder range of motion of the patients is evaluated in abduction, flexion, and external rotation. Higher measurements represent a better outcome
Change in Quick The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire score | 3 months
  The Quick DASH is an 11-item measure of the magnitude of disability and symptoms specific to the upper extremity. The first 6 items measure the degree of difficulty in performing various physical activities because of a shoulder, arm, and hand problem, and the other 5 items related to quality of sleeping, social activities, and daily activities, and the intensity of pain and numbness.
Change in Fugl-Meyer Assessment score | 3 months
  The FM scale is a 226-point multi-item Likert-type scale developed as an evaluative measure of recovery from hemiplegic stroke. It is divided into 5 domains: motor function, sensory function, balance, joint range of motion, and joint pain. Each domain contains multiple items, each scored on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully).

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Bagcier, Principal Investigator — Kars State Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Kars State Hosital, Kars
  - Kars State Hospital, Kars

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared upon reasonable request

REFERENCES:
- [Derived] Bagcier F, Yurdakul OV, Deniz G, Akbulut A, Celik Y, Temel MH. Is Dry Needling Treatment an Extra Contribution to Conventional Treatment for Hemiplegic Shoulder Pain? A Prospective, Randomized Controlled Study. Med Acupunct. 2023 Oct 1;35(5):236-245. doi: 10.1089/acu.2023.0060. Epub 2023 Oct 17. PMID 37900876